CLINICAL TRIAL: NCT04080895
Title: A Randomized, Open-Label Study to Evaluate Potential Pharmacokinetic Interactions of Orally Administered Artemether-lumefantrine and Amodiaquine in Healthy Adult Subjects
Brief Title: Pharmacokinetic Study of Artemether-lumefantrine and Amodiaquine in Healthy Subjects
Acronym: ALAQ
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was made due to the expired investigational drug and regulatory changes by the Thai FDA, along with increased importation costs. The research team and investigational drug sponsor agreed to seek approval for early project termination.
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAL19003
Record Dates: First submitted 2019-06-10; First posted 2019-09-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-04

CONDITIONS: Pharmacokinetic; Healthy; Drug Combination
Keywords: Artemether-lumefantrine; Amodiaquine
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; Amodiaquine

STUDY DESIGN:
Intervention Model Description: This is an open-label pharmacokinetic study in 16 healthy Thai subjects. Subjects will be admitted in the inpatient ward and will be randomized to group A or group B to receive 3 drug regimens (Regimen 1 Artemether-lumefantrine; Regimen 2 Amodiaquine ; Regimen 3 Artemether-lumefantrine + Amodiaquine) on Day 0, 1, and 2. Every subject will have 1 screening and 3 admissions in the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental)
  Interventions: Drug: Artemether-lumefantrine; Drug: Amodiaquine; Drug: Artemether-lumefantrine + Amodiaquine
- group B (Experimental)
  Interventions: Drug: Amodiaquine; Drug: Artemether-lumefantrine; Drug: Artemether-lumefantrine + Amodiaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Artemether-lumefantrine on Day 0, 1 and 2 Washout period: more than 6 weeks
  Arms: group A
Drug: Amodiaquine — Amodiaquine on Day 0, 1 and 2 Washout period: more than 6 weeks
Drug: Artemether-lumefantrine — Artemether-lumefantrine on Day 0, 1 and 2 Washout period: more than 6 weeks
  Arms: group B
Drug: Artemether-lumefantrine + Amodiaquine — Artemether-lumefantrine + Amodiaquine on Day 0, 1 and 2

SUMMARY:
This is an open-label pharmacokinetic study in 16 healthy Thai subjects. To assess the safety and tolerability and pharmacological interactions of the combination of artemether-lumefantrine and amodiaquine.

This study is funded by Prof White's WT PRF. The Welcome Trust grant reference number is B9R04920.

DETAILED DESCRIPTION:
This study will enroll 16 healthy subjects both male and female, aged 18-60 years, at the Clinical Therapeutic Unit, Faculty of Tropical Medicine, Mahidol University. Subjects will be healthy HIV-1, hepatitis B and C uninfected individuals who comprehend the purpose of the study and have provided written consent. All subjects will undergo screening assessments (visit 1). Screening assessments (visit 1) may be carried out over more than one day, provided that all required assessments are completed within the 14 days prior to visit 2. If the interval between screening (visit 1) and day -1 visit 2 is three days or less, the clinical laboratory screening test result and serum pregnancy test result can be used for enrolment evaluation on day -1 visit 2. In such cases, these tests would not need to be repeated at day-1 visit 2.

Visit 1 (Screening visit): All laboratory assessments (chemistry, hematology, FBS and urinalysis) must be drawn in the fasting state (8 hours fast) including serum pregnancy testing (if appropriate)

Visit 2-4: 16 healthy subjects who fulfill the eligibility criteria will be recruited and randomized to the study. All laboratory assessments (chemistry, hematology, FBS and urinalysis) must be drawn in the fasting state (8 hours fast). Results of these tests are to be available and reviewed prior to each subject receiving the study drug on day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Male or female non-smoker aged between 18 years to 60 years.
3. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and agrees to abstain from sexual intercourse or use effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
4. A male is eligible to enter and participate in this study if he: agrees to abstain from sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
5. Normal electrocardiogram (ECG) with QTc <450 msec.
6. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes (heart failure, hypokalemia) or with a family history of long QT syndrome, Brugada syndrome, or sudden cardiac death.
5. Abnormal serum creatinine (Scr) and estimated glomerular filtration rate (eGFR) <70 mL/min as determined by CKD-EPI equation
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 x half-life, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. AST or ALT >1.5 times the upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. Abnormal methemoglobin level (more than 3 mg/dL).
16. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 6 months.
17. Subject who have received quinacrine in last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC0-∞) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.
Area under the concentration-time curve AUC (0-last) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.
maximum concentration (Cmax) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.

SECONDARY OUTCOMES:
Elimination clearance (CL/F) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.
terminal elimination half-life (t1/2) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.
apparent volume of distribution (Vd) | approximately 6 - 12 months
  of artemether, lumefantrine and amodiaquine and their metabolites when given alone and in combination.
Number of adverse events | approximately 6 - 12 months
  Adverse events will be assessed as one of safety and tolerability parameters.
Number of event concerning of abnormal electrocardiograph | approximately 6 - 12 months
  Electrocardiographic changes especially QTc interval prolongation will be assessed as one of safety and tolerability parameters.
Number of event concerning of abnormal vital signs | approximately 6 - 12 months
  Abnormal vital signs will be assessed as one of safety and tolerability parameters.
Number of event concerning of abnormal laboratory values | approximately 6 - 12 months
  Abnormal laboratory values will be assessed as one of safety and tolerability parameters.
Pharmacogenetic polymorphisms identification | approximately 6 - 12 months
  Genotyping will be performed to identify polymorphisms of cytochrome 450 and other enzymes related to drug metabolism from subject who is an unusual metabolizer.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With subject's consent, subject's clinical data and results from blood analyses stored in our database may be shared with other researchers to use in the future.

DOCUMENTS (2):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04080895/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04080895/SAP_003.pdf